CLINICAL TRIAL: NCT04845555
Title: Association Between Individual Clotting Factor Level Monitoring and the Risk of Bleeding Whilst Physical Active Conditions
Acronym: AIM-Active
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prof. Dr. Dr. Thomas Hilberg (Other)
Collaborators: Takeda (Industry); University of Bonn (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Dr. Thomas Hilberg, Prof. Dr. med. Dr. phil., University of Wuppertal
Organization: University of Wuppertal (Other)
Other Study IDs: 002286
Record Dates: First submitted 2020-07-28; First posted 2021-04-15 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Clotting Factor Level; Exercise; Pharmacokinetics; Physical activity
MeSH Terms: conditions — Hemophilia A; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hemophilia A: Patients suffering from moderate or severe hemophilia A (FVIII <5%) over the age of 12 years.
  Interventions: Other: Observation of the association between clotting factor level and risk of bleeding whilst physical activity

INTERVENTIONS:
Other: Observation of the association between clotting factor level and risk of bleeding whilst physical activity — The participants of this study will be monitored for a period of twelve months regarding individual clotting factor level, bleeding episodes as well as type and intensity of physical activity. By doing so, bleeding events, factor consumption as well as the course of the individual factor clotting factor level will be documented via the mobile application "myPKFiT". This individual factor treatment regime will be compared with the retrospective treatment outcome in the last twelve months before the first study visit.

SUMMARY:
The aim of this prospective multicentre study is to evaluate the influence of individual clotting factor level while being physically active

DETAILED DESCRIPTION:
In patients with haemophilia (PwH) repetitive joint bleedings result in a so called haemophilic arthropathy, which is often associated with chronic pain as well as functional restrictions.

Due to the opportunity of sufficient factor treatment regimes, physical activity is no longer considered as a risk factor for PwH. In contrast, the large amount of current scientific evidence demonstrated high benefits of regular exercising for PwH. Meanwhile, physical activity is integrated as recommendation in the ´Guidelines for the management of hemophilia´. Nevertheless, the detailed influence of the exact course of the individual clotting factor level corresponding to the intensity of physical activities in consideration of possible bleeding events in adult PwH have not been examined to date.

The aim of this prospective multicentre study is to evaluate the influence of individual clotting factor level while being physically activie. Hereby the focus is on haemophilic specific parameters such as bleeding events, factor treatment and pain. On the basis of this study, an individualized clotting factor level should be determined which ensures a minimized risk of a bleeding event, considering type and intensity of the exercises. In line with these new findings, further interventional studies could be initiated in order to safely enhance the degraded physical performance as well as quality of life in PwH.

The generated knowledge could be further used in the development of haemophilic specific recommendations regarding physical activity in consideration of the individual clotting factor level.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from moderate or severe hemophilia A (FVIII <5%, ≥ 12 years old)
* factor treatment with ADVATE© or ADYNOVI©
* use of myPKFiT

Exclusion Criteria:

* patients suffering from other coagulopathies
* participants without written consent
* participants < 12 years old
* joint surgery like arthroscopy, synovectomy up to six months before study
* suffering from different rheumatologic diseases like M. Bechterew, Psoriasi or other local or generalized joint infections (Borreliosis, septic arthritis)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from hemophilia A recruited by cooperating hemophilic treatment centers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Type of physical activity documented in a digital template | 12 months
  PwH are used to document the type and intensity of their physical activity in terms of a digital template which will be electronically requested monthly by co-workers of this study
Physiological parameters (heart rate of PwH, measured with FitBit Charge 4 HR) | 12 months
  Individual type and intensity of physical activity measured as heart rate by an electronic activity wristband (Fitbit charge 4 HR, synchronized in corresponding FitBit Application) For the final evaluation, each physical activity will be clustered regarding type and intensity to differ between the specific demands of activity.
Total annual bleeding rate | 12 months
  Number of bleedings per year, documented in a digital template
Clotting factor VIII level | 12 months
  In percent, documented in "myPKFIT"

SECONDARY OUTCOMES:
Factor substitution in international units | 12 months
  Administered international units of factor VIII
Frequency of factor substitution | 12 months
  Frequency and units of factor replacement
Score of subjective quality of life measured by the SF36 Health Survey | Baseline, after 6 and 12 months
  Questionnaire: The possible score ranges from 0 to 100 points. 0 points represent the greatest possible restriction of health, while 100 points represent the absence of health restrictions
Joint status in score points measured by Hemophilia Joint Health Score | Baseline, after 6 and 12 months
  The clinical joint situation will be examined in all PwH and controls by the Haemophilia Joint Health Score, which assesses, e.g., swelling, muscle atrophy, crepitus on motion, axial deformity and range of motion. Higher score points imply an increased deficit in the functional and structural joint status as a sign of more pronounced haemophilic arthropathy, with a maximum possible value of 26 score points for knee and ankle joints and a maximum of 20 score points for elbow joints
Pain status measured by the German Pain Questionnaire | Baseline, after 6 and 12 months
  Questionnaire includes: Demographic data (age, sex, body weight, height); detailed subjective description of pain (localization, characteristics, time course, intensity, etc.); assessment of pain-relieving and pain-enhancing conditions, subjective pain perception (the pain description list SBL); pain-related impairment (also valid for Von Korff grading); subjective pain model, causal attribution, relieving or enhancing factors; screening of depressive and anxiety disorders (Depression, Anxiety and Stress Scale, DASS). Screening of depressive and anxious disorders (Depression, Anxiety and Stress Scale, DASS); General well-being (Marburg Questionnaire on Habitual Well-being, MFHW); Course of disease (extent of previous treatment, physicians consulted for pain, use of medication, pain therapy treatment procedures, operations); Medical and psychological/psychiatric comorbidity
Pressure pain thresholds | Baseline, after 6 and 12 months
  Pressure pain thresholds will be examined by using a digital algometer device (FPX 25 Compact Digital Algom-eter, Wagner Instruments, Greenwich, CT, USA) with a robe area of 1 cm2. Pressure is increased by a rate of 10 Newton/second. It is a measuring method to analyze the current pain condition. Participants are instructed to report the moment when the stimulus becomes painful for the first time. The maximum pressure is 140 N to avoid tissue damages. The mean value of three measurements will be used as pressure pain thresholds for further statistical analyses. Pressure pain thresholds of knee, ankle, elbow, sternum and forehead (the last two being the reference points) will be examined.
Score of subjective physical performance measured by the HEP-Test-Q | Baseline, after 6 and 12 months
  Questionnaire of subjective physical functioning for patients with hemophilia.The HEP Test-Q consists of 25 items belonging to 4 dimensions 'flexibility', 'strength & coordination', 'endurance' and 'body perception' and a single item that measures changes in physical functioning compared to the previous year. Subscales and total score are transformed to a 0-100 scale, with high scores representing better physical functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hilberg, Prof., Study Chair — Head of Department of sports medicine Wuppertal
Locations (1):
- Department of Sports Medicine, University of Wuppertal, Wuppertal, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No